CLINICAL TRIAL: NCT02877004
Title: A Feasibility Study Addressing the Frequency of Low Level Laser Therapy for Reducing Central Adiposity and Weight in Overweight Individuals
Brief Title: LLLT for Reducing Waste Circumference and Weight
Acronym: LLLT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Ivana Croghan, Professor, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16-004817
Record Dates: First submitted 2016-08-17; First posted 2016-08-24 (Estimated); Results first posted 2019-09-13 (Actual); Last update posted 2019-09-13 (Actual); Status verified 2019-09

CONDITIONS: Weight Loss
MeSH Terms: conditions — Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Laser for 4 weeks (Active Comparator): 3 Low-Level Laser Therapy Treatments Weekly
  Interventions: Device: 3 Low-Level Laser Therapy Treatments Weekly
- Laser for 6 weeks (Active Comparator): 2 Low-Level Laser Therapy Treatments Weekly
  Interventions: Device: 2 Low-Level Laser Therapy Treatments Weekly
- Laser for 12 weeks (Active Comparator): 1 Low-Level Laser Therapy Treatment Weekly
  Interventions: Device: 1 Low-Level Laser Therapy Treatment Weekly

INTERVENTIONS:
Device: 3 Low-Level Laser Therapy Treatments Weekly — Receives 12 LLLT treatment - at a frequency of 3 times per week for 4 weeks
  Arms: Laser for 4 weeks
Device: 2 Low-Level Laser Therapy Treatments Weekly — Receives 12 LLLT treatments - at a frequency of 2 times per week for 6 weeks
  Arms: Laser for 6 weeks
Device: 1 Low-Level Laser Therapy Treatment Weekly — Receive 12 LLLT treatments - at a frequency of once per week for 12 weeks
  Arms: Laser for 12 weeks

SUMMARY:
The purpose of this research is to gather preliminary information on the effectiveness of Low Level Laser Therapy (LLLT) in helping people reduce their weight gain in the central body region.

DETAILED DESCRIPTION:
This will be an open label clinical trial with all study participants receiving LLLT. Preliminary data will be collected on the efficacy of LLLT based on varying frequency of treatments. The focus of this study on 60 overweight adults with a BMI of 25 to 29.9, and assess changes in weight and waist circumference at end of treatment for group 1 (week 4) and group 2 (week 6) and group 3 (week 12). Participants will be randomized to receive LLLT treatments either 3 times a week; 2 times a week; or once a week.

ELIGIBILITY:
Inclusion Criteria:

1. over 18 years of age;
2. body weight of greater than 50 kg (110 pounds);
3. BMI between 25-29.9 kg/m2;
4. able to participate fully in all aspects of the study
5. understood and signed study informed consent

Exclusion Criteria:

1. used weight loss medications or participated in a weight loss program within past 30 days
2. currently taking supplements known to affect weight (garcinia cambogia, etc.)
3. weight fluctuations of 20 pounds or more in the past 6 months
4. implanted device (including pacemaker or lap band) in the targeted area of LLLT
5. known active eating disorder
6. known, active, untreated clinically significant psychiatric condition (alcohol or substance abuse, psychosis, bipolar disorder, or depression)
7. used an investigational drug within 30 days of study enrollment
8. currently pregnant or lactating, or are of child-bearing potential or are likely to become pregnant during the medication phase and unwilling to use a reliable form of contraception
9. history of any major cardiovascular events
10. current uncontrolled hypertension
11. clinically significant acute or chronic progressive or unstable neurologic, hepatic, renal, cardiovascular, lymphatic, respiratory, or metabolic disease
12. Prior surgical intervention for body sculpting/weight loss
13. medical, physical, or other contraindications for body sculpting/weight loss
14. any medical condition known to affect weight levels or to cause bloating or swelling
15. diagnosis of, and/or taking medication for, irritable bowel syndrome
16. active infection, wound or other external trauma to the areas to be treated with the laser
17. known photosensitivity disorder;
18. current active cancer or currently receiving treatment for or within 1 year of cancer remission

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-09-30 (Actual); Primary Completion 2018-07-28 (Actual); Study Completion 2018-08-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ivana T Croghan, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Croghan IT, Hurt RT, Schroeder DR, Fokken SC, Jensen MD, Clark MM, Ebbert JO. Low-level laser therapy for weight reduction: a randomized pilot study. Lasers Med Sci. 2020 Apr;35(3):663-675. doi: 10.1007/s10103-019-02867-5. Epub 2019 Aug 31. PMID 31473867

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants recruited from the local community of Rochester, MN, 09/16-08/17. All interested individuals called a central number and underwent a 10-minute phone pre-screen. If they passed the telephone pre-screen, they were invited to attend an in-person consent visit. All study visits and treatments took place in Mayo Clinic - Rochester Campus.
Pre-assignment Details: After consent, patients were screened for study entry criteria. Only those who passed all criteria were invited to be randomized to study.
Period: Overall Study
Arm/Group | Laser for 4 Weeks | Laser for 6 Weeks | Laser for 12 Weeks
Started | 20 | 20 | 20
Completed | 20 | 20 | 19
Not Completed | 0 | 0 | 1
Not completed — Pregnancy | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Laser for 4 Weeks | Laser for 6 Weeks | Laser for 12 Weeks | Total
Number analyzed (Participants) | 20 | 20 | 20 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 20 | 20 | 19 | 59
  >=65 years | 0 | 0 | 1 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.6 (8.3) | 40.8 (8.7) | 45.8 (10.1) | 43.7 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 20 | 19 | 54
  Male | 5 | 0 | 1 | 6
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: White/Non Hispanic | 18 | 20 | 19 | 57
  Race/Ethnicity: Other | 2 | 0 | 1 | 3
Weight (kg) [Mean (Standard Deviation); unit: Kg] | 81.7 (10.5) | 77.1 (6.8) | 75.4 (7.9) | 78.1 (8.8)
Waist Circumference (cm) [Mean (Standard Deviation); unit: cm] | 93.2 (7.0) | 91.4 (7.2) | 91.2 (6.5) | 91.9 (6.9)

OUTCOME MEASURES:

1. Primary Outcome: Change in Weight
Description: Comparison of weight change from baseline between arms
Time Frame: baseline and 4 weeks
Measure: Mean (Standard Deviation); unit: Kg
Arm/Group | Laser for 4 Weeks | Laser for 6 Weeks | Laser for 12 Weeks
Number analyzed (Participants) | 20 | 20 | 20
Kg | -0.5 (1.7) | -0.9 (1.7) | -0.6 (1.5)
Statistical Analysis 1: Comparison: Laser for 4 Weeks vs Laser for 6 Weeks vs Laser for 12 Weeks; Test type: Superiority; p = 0.723, ANCOVA; Data were analyzed using analysis of covariance with the baseline value included as the covariate

2. Primary Outcome: Change in Waist Circumference
Description: Comparison of waist circumference change from baseline between arms
Time Frame: baseline and 4 weeks
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Laser for 4 Weeks | Laser for 6 Weeks | Laser for 12 Weeks
Number analyzed (Participants) | 20 | 20 | 20
cm | -1.4 (2.3) | -2.0 (2.5) | -0.8 (2.6)
Statistical Analysis 1: Comparison: Laser for 4 Weeks vs Laser for 6 Weeks vs Laser for 12 Weeks; Test type: Superiority; p = .368, ANCOVA; Data were analyzed using analysis of covariance with the baseline value included as the covariate

ADVERSE EVENTS:
Time Frame: Adverse events were collected during LLLT treatment for each group (4 weeks for group A; 6 weeks for group B; 12 weeks for group C).
Description: All Adverse Events that met criteria for being Serious Adverse Events were recorded and followed up; In addition, adverse events not meeting SAE criteria and considered to be potentially related to the LLLT were also documented.
Arm/Group | Laser for 4 Weeks | Laser for 6 Weeks | Laser for 12 Weeks
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 1/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Laser for 4 Weeks (N=20) | Laser for 6 Weeks (N=20) | Laser for 12 Weeks (N=20)
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1) — Pregnancy - not considered related to treatment

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-10-28): https://cdn.clinicaltrials.gov/large-docs/04/NCT02877004/Prot_SAP_000.pdf